CLINICAL TRIAL: NCT03995277
Title: Investigator-Initiated Study to Evaluate the Effect of Biotin Ingestion On Routine Laboratory Tests
Brief Title: Effect of Biotin on Routine Laboratory Values
Acronym: SafeLab-HAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. med. Mahir Karakas (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Mahir Karakas, Coordinating Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: SafeLab
Record Dates: First submitted 2019-06-17; First posted 2019-06-24 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Biotin Ingestion; Interference With Routine Analyical Tests
Keywords: Biotin
MeSH Terms: interventions — Biotin

STUDY DESIGN:
Intervention Model Description: Participants take 10 mg/d of biotin at the same time each morning for 10 days. Blood draw for biobanking will be collected at baseline prior to starting biotin (day 1), after 10 days of biotin supplementation (day 10), and 10 days after participants stopped taking biotin (day 20).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy cohort - high dose (Other): Apparently healthy subjects, who take 10 mg/d of biotin at the same time each morning for 10 days. Blood draw for biobanking will be collected at baseline prior to starting biotin (day 1), after 10 days of biotin supplementation (day 10), and 10 days after participants stopped taking biotin (day 20).
  Interventions: Dietary Supplement: Biotin
- Hypothyroid cohort (Other): Subjects under thyroid medication, who take 10 mg/d of biotin at the same time each morning for 10 days. Blood draw for biobanking will be collected at baseline prior to starting biotin (day 1), after 10 days of biotin supplementation (day 10), and 10 days after participants stopped taking biotin (day 20).
  Interventions: Dietary Supplement: Biotin
- Healthy cohort - low dose (Other): Apparently healthy subjects, who take 50 µg/d of biotin at the same time each morning for 20 days. Blood draw for biobanking will be collected at baseline prior to starting biotin (day 1), after 10 days of biotin supplementation (day 10), after 20 days of biotin supplementation (day 20), and 10 days after participants stopped taking biotin (day 30).
  Interventions: Dietary Supplement: Biotin

INTERVENTIONS:
Dietary Supplement: Biotin — Daily intake of 10 mg or 50 µg per day

SUMMARY:
Inaccuracy of laboratory medicine diagnostic tests may be associated with ingestion of over-the-counter biotin supplements.

DETAILED DESCRIPTION:
Study group 1) Due to a lack of systematic studies, little is known about how performance of specific biotinylated immunoassays is associated with biotin ingestion at doses common in over-the-counter supplements (10 mg/d) in healthy adults and subjects with thyroid hormone supplementation. Therefore, this study was designed to assess the association of short-term biotin ingestion for 10 days with performance of various analytes based on Roche, Abbott and Siemens assays.

Study group 2) Due to a lack of systematic studies, little is known about how performance of specific biotinylated immunoassays is associated with biotin ingestion at doses common in multivitamin supplements (biotin = 50 µg/d) in healthy adults. Therefore, this study was designed to assess the association of short-term biotin ingestion for 20 days with performance of various analytes based on Roche, Abbott and Siemens assays.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Apparently healthy

Exclusion Criteria:

* Pre-existing condition other than hypothyroidism
* Intake of dietary supplements containing biotin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Variance of routine analyte concentrations | 20 days (high-dose groups) and 30 days (low-dose group)
  The study aims to assess the performance of specific biotinylated immunoassays after 10 days of ingesting 10 mg/d of biotin (high-dose), or 50 µg/d of biotin (low-dose). Control measurements will be performed at baseline (before biotin intake), and 10 days after last biotin intake.

CONTACTS AND LOCATIONS:
Overall Officials: Mahir Karakas, MD, MBA, Principal Investigator — University Heart Center Hamburg
Locations (4):
- Germany (4):
  - University of Augsburg, Augsburg
  - University Heart Center Hamburg, Hamburg
  - University of Hamburg, Hamburg
  - University of Mainz, Mainz

IPD SHARING:
Plan to Share IPD: Undecided